CLINICAL TRIAL: NCT07039305
Title: Modified Cardiac Rehabilitation to Enhance Post-Stroke Physical and Psychosocial Function: Does Depression Limit the Response?
Brief Title: Physical Capacity Building for Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Ryan Ross, Assistant Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00140518; R01HD114673 (NIH)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Post-stroke Depression
Keywords: Depression; Exercise; Stroke; Stroke Recovery
MeSH Terms: conditions — Stroke; Depression; Motor Activity | interventions — Muscle Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Physical capacity training (Experimental): Physical capacity training is a comprehensive modified cardiac rehabilitation program consisting of aerobic and resistance exercise. Participants will attend a total of 36 sessions of training.
  Interventions: Behavioral: Physical capacity training for chronic stroke - building aerobic capacity and muscle strength

INTERVENTIONS:
Behavioral: Physical capacity training for chronic stroke - building aerobic capacity and muscle strength — The general format of each exercise session includes assessment of resting heart rate (HR), blood pressure (BP), and rating of perceived exertion (RPE) followed by a 5-minute warm-up, a minimum of 30 minutes of aerobic exercise followed by 25 minutes of resistance exercise. Aerobic exercise will always include a minimum of 10 minutes of walking (overground or treadmill) at the prescribed intensity followed by cycle, arm or rowing ergometry. Sessions will begin at a target intensity of ~60% heart rate reserve (HRR) determined from the exercise tolerance test performed at baseline and calculated using Karvonen's formula. The goal will be to increase training intensity by ~5% HRR every ~3 weeks and progressed as tolerated. Resistance exercise will target all major muscle groups and include multiple sets dosed at the 10-repetition to fatigue level (~75% of the 1-repetition maximum). Resistance exercises will be progressed with improvements in strength or as tolerated.

SUMMARY:
Cardiac rehabilitation is the standard-of-care treatment option for patients with cardiovascular disease and has been shown to improve many aspects critical to patient recovery. Investigators believe that individuals who have had a stroke need to be treated similarly. Investigators will study the effects of a comprehensive modified cardiac rehabilitation program to determine if it can improve some of the physical and psychosocial problems common in survivors of stroke with and without depression.

DETAILED DESCRIPTION:
Cardiac rehabilitation is a mandated, standard-of-care treatment for patients following cardiac events (e.g., heart attack, angioplasty, cardiac bypass). Cardiac rehabilitation is designed to enhance recovery via progressive exercise and is shown to improve overall physical, cognitive and psychosocial function. Disappointingly, despite sharing common etiology and post-event risk factors, stroke is not a condition that qualifies survivors for cardiac rehabilitation and few clinical trials that have directly investigated the impact of a comprehensive modified cardiac rehabilitation program on physical and psychosocial function in chronic survivors of stroke. Moreover, depression is the most common neuropsychiatric manifestation following stroke, and subjects with post-stroke depression (PSD) are historically excluded from rehabilitation clinical trials. Consequently, data describing the effects of a cardiac rehabilitation programs on physical and psychosocial function in cohorts with PSD is lacking. The purpose of this project is to examine the effects of Physical Capacity training for ChroniC stroke - Building Aerobic capacity and Muscle Strength (PC3-BAMS), a 12-week modified cardiac rehabilitation program, on physical and psychosocial function in community-dwelling survivors of stroke with and without post-stroke depression (PSD).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* A diagnosis of stroke at least 6 months prior
* Residual paresis in the lower extremity (Fugl-Meyer lower extremity [LE] motor score <34)
* Ability to walk without assistance and without an AFO during testing and training at speeds ranging from 0.2-1.0 m/s
* Ability to follow instructions, complete cognitive testing and to communicate exertion, pain and distress
* No antidepressant medications or no change in doses of psychotropic medication for at least 4 weeks prior to the study (6 weeks if newly initiated medication)
* HDRS17 question #3 and PHQ-9 question #9 regarding suicide ≤ 2
* Provision of informed consent.

In addition, depressed subjects will screen for probable major depressive disorder (Patient Health Questionnaire-9 ≥ 10) and be diagnosed using the Structured Clinical Interview for Depression (SCID) according to the DSM-5.

Exclusion Criteria:

* Unable to ambulate at least 150 feet or experienced intermittent claudication while walking
* Unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during ADL's
* Dementia
* Life expectancy <1 yr
* History of DVT or pulmonary embolism within 6 months
* Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions
* Severe hypertension with systolic >200 mmHg and diastolic >110 mmHg at rest
* Attempt of suicide in the last 2 years or suicidal risk assessed by depression screening
* Current enrollment in a rehabilitation trial to enhance motor, cognitive and or psychosocial recovery
* Severe cognitive impairment (MoCA score ≤15)
* Moderate to severe neglect that precludes cognitive testing

For brain stimulation procedures only:

* Electronic or metallic implants
* History of seizures
* Women of child bearing potential

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test | From enrollment to the end of treatment at 12 weeks
  Distance walked in six minutes.
Stroke Impact Scale | From enrollment to the end of treatment at 12 weeks
  The SIS assesses post-stroke recovery across eight domains - social participation, emotion, communication, memory, mobility, strength, hand function, and activities of daily living - as well as subjective extent of overall recovery.
Hamilton Depression Rating Scale - 17 | From enrollment to the end of treatment at 12 weeks
  The Hamilton Depression Rating Scale interview contains 17 items that assess the severity and frequency of depressive symptoms over the previous week.

SECONDARY OUTCOMES:
Peak aerobic capacity | From enrollment to the end of treatment at 12 weeks
  Peak aerobic capacity will be determined from a standardized cardiopulmonary exercise test and collection of expired gases.
Inventory of Psychosocial Functioning | From enrollment to the end of treatment at 12 weeks
  The Inventory of Psychosocial Functioning is an 80-item measure that assesses perceived frequency of function across multiple domains of life including romantic relationships, family other than spouse/partner, work, friendships and socializing, parenting, education, and self-care.
Self-selected walking speed | From enrollment to the end of treatment at 12 weeks
  Self-selected walking speed will be assessed on an instrumented mat that measures spatiotemporal characteristics of walking.

OTHER OUTCOMES:
Brain-derived neurotrophic factor | From enrollment to the end of treatment at 12 weeks
  Resting concentrations of serum and plasma brain-derived neurotrophic factor will be assessed through blood specimen collections.
Corticomotor plasticity | From enrollment to the end of treatment at 12 weeks
  Corticomotor plasticity will be assessed using a non-invasive brain stimulation paradigm called paired associative stimulation (PAS). PAS utilizes a repeated and timed peripheral nerve stimulation combined with transcranial magnetic stimulation (TMS) of the contralateral motor cortex to assess corticomotor plasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Ross, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, physical function, psychosocial function, and physiological data will be collected. Study data will be captured in a secure electronic data capture system and submitted to the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH) after all 18 HIPAA identifiers have been removed. The original dataset will be preserved at the Principal Investigator's institution. The sample informed consent, protocol, data collection forms, standardized assessment forms, data dictionary, and code book will be available in NICHD-DASH. We will use the DASH Codebook to guide our submission of variable-level metadata. The DASH codebook is a templated data dictionary, and will include details of Common Data Elements, definitions, and standards used for data collection and sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study team will submit processed and cleaned data to DASH as soon as possible, and no later than the time of an associated publication or end of the performance period, whichever comes first. Data will be preserved for as long as possible within the repository's data storage and retention policies.
Access Criteria: Prior to submission of any shared data to DASH, the Medical University of South Carolina Institutional Review Board will certify that our plan for data sharing is consistent with our informed consent procedures and does not unduly increase the risk of participants being identified.
  Study data will be shared with controlled access in DASH for general research use, as allowed by the participant's informed consent and the Institutional Certification.